CLINICAL TRIAL: NCT03037190
Title: Investigation Whether a Gluten Free Diet After the Onset of Type 1 Diabetes (T1D) Can Better Preserve the Remaining Beta Cell Mass and at the Same Time Prevent the Development of Celiac Disease (CD) in These Patients.
Brief Title: Preservation of Residual Beta Cell Mass and Prevention of Celiac Disease in Children With Recent Onset Type 1 Diabetes
Acronym: Diabglut
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Annelie Carlsson, Associate Professor, Lund University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LUDU
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 1; Remission; Celiac Disease in Children
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: •The trial is designed as a 2-arm not randomized, open, multicentre study comparing 1 year of gluten free diet with normal diet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A:withdrawal of gluten from the diet, Group A will have a gluten free diet for a year after the onset of diabetes
  Interventions: Other: withdrawal of gluten from the diet
- B normal diet (No Intervention): Group B will have normal not glutenfree diet, no planned intervention

INTERVENTIONS:
Other: withdrawal of gluten from the diet — Gluten free diet the same recommendations as for patients with diabetes and known celiac disease
  Arms: Group A

SUMMARY:
The overall aim of this project is to investigate whether a gluten free diet after the onset of type 1 diabetes (T1D) can better preserve the remaining beta cell mass and at the same time prevent the development of Celiac Disease (CD) in these patients.

Specific aims

• To study whether gluten free diet during one year after the onset of diabetes influence the appearance and duration of clinical remission in children with Type 1 diabetes.

New data show that a gluten free diet is beneficial concerning the insulin production after the onset of diabetes. The investigators want to investigate if gluten is a triggering protein for the destruction of the beta cell function after the onset of diabetes by comparing children who have a normal diet compared to children with a gluten free diet during one year after the onset of the disease.

* To study whether a gluten free diet during one year after the onset of diabetes prevent the development of Celiac Disease in these children and the impact of having two diseases It is known that it is almost 10 times more common that children with Type 1 Diabetes (IDDM) develop Celiac Disease (CD) than the general population and that most of these children (6-7 %) develop CD after the onset of Diabetes and within 5 years. Based on our new data that CD is preventable to some extent the investigators plan to perform randomized controlled studies if it is possible to prevent or postpone CD by means after the onset of IDDM.
* To investigate the impact of gluten free diet on the regulation of autoimmune responses The investigators will test the hypothesis that gluten free diet in children with recent onset T1D will implement immune regulation and inhibit the activation of potentially autoreactive T cells.

DETAILED DESCRIPTION:
General project outline Our aim is to perform a intervention study whether one year gluten free diet in children with newly diagnosed TID would make it possible to influence the speed of the beta-cells destruction and if this diet decrease the risk to develop CD after the disease A power calculation shows that we would need 600 participants to detect clinically relevant effects (see power calculation). As the power calculation is based on estimated effects we plan to first perform a pilot study including 100 patients. Based on the results of the pilot study we then plan to continue to design a larger study to get more robust information.

All children will also at the start study and, after 1 and 2 years receive a KID-screen form to study the quality of life of time in children with diabetes and to compare children with diabetes without CD and to them who will develop or have undiagnosed CD. Furthermore all children will also be monitored by a dietician during the study period, at onset, after 1 and 2 years according to the content (protein, fat, carbohydrate, gluten and vitamins) during the study.

Population Consecutive patients with recent onset of diabetes at Swedish paediatric clinics are given information about the study and they and their parents are asked to participate in the trial.

Informed consent given by patients and guardians/parents and inclusion criteria are; 1. Type 1 diabetes according to the ADA classification with < 1 months diabetes duration at time of screening 2. Age 3.00 -17.99 years at time of screening 3. Fasting C-peptide at time of screening ≥ 0.12 nmol/L Exclusion Criteria

1. Inability or unwillingness to comply with the provisions of this protocol
2. Deemed by the investigator not being able to follow instructions and/or follow the study protocol Recruitment and Screening Eligible subjects and their parent(s) / guardian(s) will have the study explained to them, and will receive a written patient information. If, after this, the subjects agree to participate, they will personally sign and date the written informed consent form. In accordance with the Declaration of Helsinki, the investigator must explain to the patient that they have the right to withdraw from the study at any time, and that this will in no way prejudice their future treatment

Sample size, power calculation:

We are planning the study as a continuous response from independent control and experimental subjects with 1 control per experimental subject. In a similar study the response within each subject group was normally distributed with standard deviation 0,19. If the true difference in the experimental and control means is 0,05 we will need to study 250 subjects and 250 controls to be able to reject the null hypothesis that the population means of the experimental and control group are equal with a probability (power) 0,8. The Type 1 error probability associated with this test of this null hypothesis is 0,05. Recalculation of sample size is needed on a pilot study, which we have chosen to 100 subjects, 50 in each group. This field also benefit from that smaller and shorter trials are conducted to obtain initial sense of efficacy prior to undertake a fully powered study.

The risk to develop CD in the children with gluten free diet will be compared to the 8000 children in the BDD who had been followed yearly with transglutaminse autoantibodies for CD.

Study Design The trial is designed as a 2-arm not randomized, open, multicentre study comparing 1 year of gluten free diet with normal diet. In the pilot study 100 patients will be recruited at 7 sites in Sweden (and if the pilot study shows expected results we will include all 43 Swedish pediatric clinics and altogether an estimated 600 patients). The patients will not be randomized into two parallel groups as it could influence the compliance to a normal diet. Instead we will recruit group A (50 patients) during the first year and group B with 50 age and sex-matched patients during the second year. Group A will eat gluten free diet for a year after the onset of diabetes and B normal diet. Both groups will follow the same procedures according to the study visits and clinical routines in our diabetes care and follow up.

Eligibility: Patients who qualify for the study have to have a C-peptide over above 0.12 nmol/L and will be assigned with a number and this screening number together with the clinics, site number, will be used as patient identification. The patients will be assessed for eligibility at the screening visit (Visit 1) prior to the start of treatment with glutenfree diet and screened with a MMTT (mixed meal tolerance test) and fasting C-peptide levels.

The patients will be followed for a total study period of 60 months which includes not more than 6 extra visits for the study (however these visits may be combined with regular diabetes care visits though all children with diabetes use to attend outpatient clinic at least every 3 month and more often at the onset of the disease) Visit 1; 2 month within the onset, MMT and fasting C-peptide Visit 2; If eligible, randomized to group A (the first 50), contact with a dietitian, information of GFD, within 3 month from onset Visit 3; at 6 months; fasting C-peptide, immunological analyses and contact with a dietician; questionnaire and a registry (before the visit one week registry of the diet intake) Visit 4; at 12 months; MMTT fasting C-peptide, HbA1c, immunological analyses. HbA1c, immunological analyses for research, contact with a dietician; questionnaire and a registry (before the visit one week registry of the diet intake) Visit 5; at 18 months, MMTT fasting C-peptide, HbA1c, immunological analyses. HbA1c, immunological analyses, including Ttg (transglutaminse) Visit 6; at 24 months, MMTT fasting C-peptide, HbA1c, immunological analyses. HbA1c, immunological analyses, including Ttg (transglutaminse) yearly until 60 months. Questionnaire about quality of life and gluten content.

Both group A and B will have same information and visits according to the diabetes care where contacts with a dietician is mandatory, but arm A will need special information about a gluten free diet and will also have x-support according to gluten free products.

Both group A and B will be followed according to CD risk during 5 years with Ttg annually as a clinical routine.

Experimental strategy

AIM 1

* To investigate changes in beta-cell function the patients will undergo an MMTT (measuring C-peptide, 90 minute value and AUCmean 0-120 min) at basile baseline (Visit 1) to 12 and 18 months). Our research nurse will perform this test on all patients included at the different sites and the samples are analyzed at the Clinical Chemistry at SUS, Malmö.
* We will also investigate and compare the proportion of patients with a stimulated maximum C-peptide level above 0.2 nmol/L after 12 and 18 months respectively as well as fasting C-peptide, change between baseline and month 6, 12 and 18 months between the groups.
* Differences between metabolic control, Hemoglobin A1c (HbA1c), change between baseline and subsequent visits
* Hemoglobin A1c (HbA1c, marker of metabolic control)) as marker for long term hyperglycemia will be analyzed at baseline and subsequent visits in both groups. We will also study if there are differences in exogenous insulin dose per kg body weight and 24 hours, change between baseline and subsequent visits as indirect marker of beta cell insulin secretion.

AIM 2 To follow the development of gluten-induced humoral autoimmunity, IgA anti-tissue-transglutaminase autoantibodies (Ttg) will be determined in blood samples collected at the onset, before insulin therapy,, and yearly up to five year after the onset of TID. Ttg autoantibodies will be analyzed by enzyme-linked immunosorbent assay Aim 3

• To investigate the immunoregulatory effect of gluten-free diet we will perform a detailed analysis of the magnitude and the phenotype of both gliadin- and tTG-specific T cells. Quantitative analysis of antigen-specific T cells will be performed using multicolor flow cytometry and cytokine secretion Gender and ethnicity All our data will respect to gender and ethnicity is evaluated if there are any predictive factors associated: Diabetes is the autoimmune disease, which is more common in boys than girl, and the reason for this is unknown and Celiac Disease is more common in girls.

Ethical considerations In spite of a very heavy, intensive, expensive treatment many patients with TID get life-threatening serious both acute and late complications. At diagnosis many patients have some slight residual insulin secretion. As long as this is the case it is much easier to keep blood glucose stable, the incidence of hypoglycaemia decreases as well as the risk of keto-acidosis. A trial with a gluten free diet is not very complicated and it is safe but may be a burden for the children and families involved. Gluten free special products are often more expensive, few products and are often considered not so tasty but when summarizing the pros and cons, there is a clear possibility of therapeutic benefit of great importance with no risk.

Clinical implications Toward an individualized treatment: To find predictive a factors determining the remission period is important for people who develop diabetes. Every month in remission increase the quality of life, increase metabol control and thereby postpone late complications. To find triggering factors for to rate of beta-cells destruction unable us to design a more individualized treatment in respective individual. Increased remission period and decreased risk of developing Celiac Disease. Gluten free diet is a safe administer, well tolerable for the patients and the main long-term goal is to find a treatment at onset of Type 1 diabetes in young patients which is easy and safe and preserve residual insulin secretion and give the patients a better quality of life, with less acute complications and in the long run less risk of late complications. The identification of exogenous factors triggering and driving beta-cell destruction offers a potential means for intervention aimed at the prevention of T1D. Environmental modification is likely to offer the most powerful strategy for effective prevention of T1D, because such an approach can target the whole population or at least that proportion of the population carrying increased genetic disease susceptibility.

Diet is a cornerstone in the diabetes treatment and individuals with diabetes must always be much aware of the carbohydrate content in the food which limits the arena of different beverages and make life more complicated and if the individual has both IDDM and CD this is even more complicated and limit the social and quality of life. If this study could prevent some individuals to develop CD it would increase their life quality extensively.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes according to the ADA classification with < 1 months diabetes duration at time of screening
* Age 3.00 -17.99 years at time of screening
* Fasting C-peptide at time of screening ≥ 0.12 nmol/L

Exclusion Criteria:

* Inability or unwillingness to comply with the provisions of this protocol
* Deemed by the investigator not being able to follow instructions and/or follow the study protocol

NB: new ethical approval will be applied for children between 1-3 years of age

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Preservation of beta cells function | within 2years after the onset of type 1 diabetes
  Differences in c-peptide production between the Groups A and B, 12 and 18 months after the onset of diabetes.

SECONDARY OUTCOMES:
Prevention of Celiac DIsease | Five years after the onset of Diabetes
  Differencies in incidence of Celiac Disease between the two groups, after onset of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Annelie Carlsson, MD PhD, Principal Investigator — Lund University
Locations (1):
- Skanes University Hospital, Lund, Region Skane, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pastore MR, Bazzigaluppi E, Belloni C, Arcovio C, Bonifacio E, Bosi E. Six months of gluten-free diet do not influence autoantibody titers, but improve insulin secretion in subjects at high risk for type 1 diabetes. J Clin Endocrinol Metab. 2003 Jan;88(1):162-5. doi: 10.1210/jc.2002-021177. PMID 12519846
- [Background] Hummel S, Pfluger M, Hummel M, Bonifacio E, Ziegler AG. Primary dietary intervention study to reduce the risk of islet autoimmunity in children at increased risk for type 1 diabetes: the BABYDIET study. Diabetes Care. 2011 Jun;34(6):1301-5. doi: 10.2337/dc10-2456. Epub 2011 Apr 22. PMID 21515839
- [Background] Sildorf SM, Fredheim S, Svensson J, Buschard K. Remission without insulin therapy on gluten-free diet in a 6-year old boy with type 1 diabetes mellitus. BMJ Case Rep. 2012 Jun 21;2012:bcr0220125878. doi: 10.1136/bcr.02.2012.5878. PMID 22729336
- [Background] Ivarsson A, Myleus A, Norstrom F, van der Pals M, Rosen A, Hogberg L, Danielsson L, Halvarsson B, Hammarroth S, Hernell O, Karlsson E, Stenhammar L, Webb C, Sandstrom O, Carlsson A. Prevalence of childhood celiac disease and changes in infant feeding. Pediatrics. 2013 Mar;131(3):e687-94. doi: 10.1542/peds.2012-1015. Epub 2013 Feb 18. PMID 23420914